CLINICAL TRIAL: NCT00674570
Title: Effects of Hydrocortisone and D-Cycloserine on Fear Extinction in Veterans With Posttraumatic Stress Disorder
Brief Title: Veteran Stress and Learning Study
Acronym: VSL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CDA-2-037-07F; H841-31915-01A (Other: San Francisco VAMC)
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Stress Disorders, Posttraumatic
Keywords: Stress Disorders, Posttraumatic; Hydrocortisone; Cycloserine; Extinction, Psychological; PTSD; San Francisco
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Hydrocortisone; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm 1: Hydrocortisone (Experimental): Hydrocortisone
  Interventions: Drug: Hydrocortisone
- Arm 2: D-Cycloserine (Experimental): D-Cycloserine
  Interventions: Drug: D-Cycloserine
- Arm 3: Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — 25 mg/oral one hour prior to extinction task
  Arms: Arm 1: Hydrocortisone
Drug: D-Cycloserine — 50 mg/oral one hour prior to extinction task
  Arms: Arm 2: D-Cycloserine
Drug: Placebo — One hour prior to extinction task
  Arms: Arm 3: Placebo

SUMMARY:
This is a research study examining the use of two medications, Hydrocortisone and D-Cycloserine, compared to an inactive substance (placebo), on their ability to reduce fear responses and memory of fear in Veterans with symptoms of Posttraumatic Stress Disorder (PTSD). These responses will be tested using a fear learning and memory task administered by computer.

ELIGIBILITY:
Inclusion Criteria:

* Veterans and civilians with an age range of 18 to 65 years
* Participants must be physically healthy volunteers

Exclusion Criteria:

* Individuals who fall outside the age range
* Individuals with medical conditions that would interfere with participation
* Other criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2009-01-13 (Actual); Primary Completion 2015-06-22 (Actual); Study Completion 2015-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabra S Inslicht, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexandra Kredlow M, Pineles SL, Inslicht SS, Marin MF, Milad MR, Otto MW, Orr SP. Assessment of skin conductance in African American and Non-African American participants in studies of conditioned fear. Psychophysiology. 2017 Nov;54(11):1741-1754. doi: 10.1111/psyp.12909. Epub 2017 Jul 4. PMID 28675471
- [Background] Inslicht SS, Metzler TJ, Garcia NM, Pineles SL, Milad MR, Orr SP, Marmar CR, Neylan TC. Sex differences in fear conditioning in posttraumatic stress disorder. J Psychiatr Res. 2013 Jan;47(1):64-71. doi: 10.1016/j.jpsychires.2012.08.027. Epub 2012 Oct 26. PMID 23107307
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participation involved 4 study visits, with randomization to intervention arm and drug administration occurring on visit 3. The discrepancy between 111 participants who were initially enrolled and 106 at randomization resulted from 5 participants who dropped out between screening and visit 3, when they were to have been assigned into a group.
Period: Overall Study
Arm/Group | Arm 1: Hydrocortisone | Arm 2: D-Cycloserine | Arm 3: Placebo
Started (5 participants dropped out between screening and randomization to group.) | 37 | 34 | 35
Completed | 37 | 32 | 35
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Hydrocortisone | Arm 2: D-Cycloserine | Arm 3: Placebo | Total
Number analyzed (Participants) | 37 | 34 | 35 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (12.8) | 41.1 (13.7) | 40.0 (11.8) | 38.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 18 | 62
  Male | 14 | 13 | 17 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 7 | 18
  Not Hispanic or Latino | 30 | 30 | 28 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 6 | 7 | 18
  White | 22 | 21 | 25 | 68
  More than one race | 7 | 3 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 34 | 35 | 106

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Maximum Skin Conductance Response (SCR) in Microsiemens (µS)
Description: Psychophysiology measurements occurred on day 7 for fear conditioning, day 9 for fear extinction, and day 11 for extinction retention. The primary outcome measures are presented for the first and last conditioned stimulus (CS) trials during fear conditioning and extinction and for the first 2 trials during retention. Conditioned Responses (CR): An SCR score was obtained for each CS by subtracting the mean skin conductance level (SCL) in microsiemens (µS) for the 2-s interval immediately preceding CS onset from the max SC level in µS during the 8-s CS presentation. Unconditioned Response (UCR): An SCR score for the UCR was obtained by subtracting the mean SCL in µS within 6-8 s following CS offset from the max increase in SC level during the .5-6.5 time interval following the CS offset, corresponding to the onset of the .5s US. SC responses were range corrected using each participant's maximum response to the UCS or CS during acquisition trials of the fear conditioning phase.
Time Frame: 15 minute measurement intervals on Study Days 7, 9, and 16
Measure: Mean (Standard Error); unit: proportion of max SCR (µS)
Arm/Group | Arm 1: Hydrocortisone | Arm 2: D-Cycloserine | Arm 3: Placebo
Number analyzed (Participants) | 37 | 32 | 35
proportion of max SCR (µS)
  Fear Conditioning: Beginning | .0325522 (.0351212) | .0245775 (.0367306) | -.0181339 (.0328529)
  Fear Conditioning: End | .1233174 (.0351212) | .1024914 (.0367306) | .1276977 (.0328529)
  Fear Extinction: Beginning | .0298132 (.0313355) | .0674658 (.0327715) | .1104578 (.0313355)
  Fear Extinction: End | .0013351 (.0313355) | -.026853 (.0327715) | .0854075 (.0313355)
  Extinction Retention | -.0101856 (.0388043) | -.0248148 (.0405825) | .0985292 (.0393708)
Statistical Analysis 1: Comparison: Arm 2: D-Cycloserine vs Arm 3: Placebo; Fear Conditioning Beginning (first trial); Test type: Superiority; p = .66, Mixed Models Analysis; Mean Difference (Net) = -.02, 95% CI 2-sided [-.15 to .10], Standard Error of Mean .06
Statistical Analysis 2: Comparison: Arm 1: Hydrocortisone vs Arm 3: Placebo; Fear Conditioning Beginning (first trial); Test type: Superiority; p = .41, Mixed Models Analysis; Mean Difference (Net) = -.05, 95% CI 2-sided [-.17 to .07], Standard Error of Mean .06
Statistical Analysis 3: Comparison: Arm 2: D-Cycloserine vs Arm 3: Placebo; Fear Conditioning End (last trial); Test type: Superiority; p = .43, Mixed Models Analysis; Median Difference (Net) = .05, 95% CI 2-sided [-.07 to .18], Standard Error of Mean .06
Statistical Analysis 4: Comparison: Arm 1: Hydrocortisone vs Arm 3: Placebo; Fear Conditioning End (last trial); Test type: Superiority; p = .47, Mixed Models Analysis; Median Difference (Net) = .04, 95% CI 2-sided [-.07 to .17], Standard Error of Mean .06
Statistical Analysis 5: Comparison: Arm 1: Hydrocortisone vs Arm 3: Placebo; Fear Extinction Beginning (first trial); Test type: Superiority; p = .065, Mixed Models Analysis; Mean Difference (Net) = .09, 95% CI 2-sided [-.01 to .20], Standard Error of Mean .05
Statistical Analysis 6: Comparison: Arm 2: D-Cycloserine vs Arm 3: Placebo; Fear Extinction Beginning (first trial); Test type: Superiority; p = .34, Mixed Models Analysis; Mean Difference (Net) = .05, 95% CI 2-sided [-.05 to .15], Standard Error of Mean .05
Statistical Analysis 7: Comparison: Arm 2: D-Cycloserine vs Arm 3: Placebo; Extinction End (last trial); Test type: Superiority; p = .003, Mixed Models Analysis; Mean Difference (Net) = .16, 95% CI 2-sided [.06 to .26], Standard Error of Mean .05
Statistical Analysis 8: Comparison: Arm 1: Hydrocortisone vs Arm 3: Placebo; Extinction End (last trial); Test type: Superiority; p = .02, Mixed Models Analysis; Mean Difference (Net) = .12, 95% CI 2-sided [.02 to .22], Standard Error of Mean .05
Statistical Analysis 9: Comparison: Arm 2: D-Cycloserine vs Arm 3: Placebo; Extinction Retention (first 2 trials) First trials were selected as a test of extinction retention, since repeated presentations of the CS without a UCS were expected to result in additional fear extinction; Test type: Other; p = .006, Mixed Models Analysis; Mean Difference (Net) = .18, 95% CI 2-sided [.05 to .30], Standard Error of Mean .06
Statistical Analysis 10: Comparison: Arm 1: Hydrocortisone vs Arm 3: Placebo; Extinction retention; Test type: Other; p = .01, Mixed Models Analysis; Mean Difference (Net) = .16, 95% CI 2-sided [.04 to .28], Standard Error of Mean .06

ADVERSE EVENTS:
Time Frame: Approximately, one month for each participant during their enrollment in the study.
Arm/Group | Arm 1: Hydrocortisone | Arm 2: D-Cycloserine | Arm 3: Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/32 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/32 | 0/35
Other Adverse Events (participants affected / at risk) | 0/37 | 0/32 | 0/35

LIMITATIONS AND CAVEATS:
Technical difficulties rendered corrugator electromyogram data unusable for analysis. We selected skin conductance as a primary measure of sympathetic activity rather than heart rate, which has both sympathetic and parasympathetic influences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No